CLINICAL TRIAL: NCT01824667
Title: Double-blind, Placebo Controlled, Randomised, Multicentered, of Parallel Design Study to Determine the Effect of B-GOS on GI Discomfort in Healthy Adults
Brief Title: Effect of B-GOS on GI Discomfort in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clasado Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CLAS/1213
Record Dates: First submitted 2013-02-25; First posted 2013-04-05 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
MeSH Terms: interventions — maltodextrin; High Fructose Corn Syrup

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- B-GOS (Experimental): 2.75g daily for 4 weeks
  Interventions: Dietary Supplement: B-GOS
- Maltodextrin (Placebo Comparator): 2.75g daily for 4 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: B-GOS
  Other Names: Bimuno
  Arms: B-GOS
Dietary Supplement: Maltodextrin
  Other Names: corn syrup
  Arms: Maltodextrin

SUMMARY:
The aim of the study is to evaluate the effects of a new food supplement which is currently available in the market, called Bimuno® (B-GOS), on gastrointestinal discomfort (e.g. bloating, abdominal pain/cramp and flatulence) in adults who often experience these symptoms but are otherwise healthy.

About 400 volunteers will take part in this study, which will last 6 weeks (to include 4 weeks treatment and 2 weeks follow up period).

Episodes of abdominal pain or discomfort (e.g. bloating, abdominal pain/cramp and flatulence), in the absence of diseases, are commonly associated with food or drug intake or with alterations of bowel habit and vary between individuals in frequency and severity.

Some dietary ingredients are known to reduce these symptoms. We have used B-GOS previously in trials with healthy younger and older adults and we have observed a trend towards reducing abdominal bloating. However, the investigators have not tested B-GOS in healthy adults who often experience these symptoms and this is what we will investigate now.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years old.
2. Presence of bloated feeling or experiencing abdominal fullness, with or without visible distention, often in the last 12 months.
3. Ability to communicate well with the investigator and to comply with the requirements of the entire study.
4. Volunteer has given written informed consent to participate and is willing to participate in the entire study.

Exclusion Criteria:

1. History or evidence of organic disease of the gastrointestinal tract; such as tumour, irritable bowel syndrome, etc., within the previous 5 years.
2. Undergone surgical resection of any part of the bowel.
3. History of malignancy within the previous 5 years (with exception of well-treated basal cell carcinoma or in situ cervical carcinoma).
4. Received antibiotics in the previous four weeks.
5. Consumed probiotic or prebiotic preparations on a regular basis (at least 3 times per week) in the last 2 weeks.
6. Former participation in another study involving prebiotic or probiotic preparations or investigational drugs within the previous one month, or intention to use such drugs during the course of the study.
7. Severe allergy or any history of severe abnormal drug reaction, drug or alcohol abuse.
8. Regular use of any medication with exception of hormonal replacement therapy and contraception.
9. Women who are pregnant or breast-feeding.
10. Fertile women not practicing a medically-approved method of contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To determine the effect of B-GOS on GI discomfort | Participants will be followed daily for 6 weeks
  questionnaires

SECONDARY OUTCOMES:
To conduct an assessment of stools | Participants will be followed daily for 6 weeks.
  questionnaires

OTHER OUTCOMES:
To assess the effect of B-GOS on the quality of life and general well being. | beginning and end of the study
  questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Research Insights Ltd, Oxford, United Kingdom